CLINICAL TRIAL: NCT06591039
Title: A Multicenter Prospective Observational Cohort Study of Breast Cancer Based on a Breast Cancer Medical Record Database in China
Brief Title: A Multicenter Prospective Observational Cohort Based on a Breast Cancer Medical Record Database in China
Status: Recruiting | Type: Observational
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Jiong Wu, chief physician, Fudan University
Other Study IDs: ATOSSA-001
Record Dates: First submitted 2024-09-02; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Breast Neoplasms
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Procedure: The study did not involve intervention in the patient's treatment regimen — This study is based on a prospective database platform to register the occurrence, treatment and prognosis of breast cancer in China, so there is no clear exposure factor. This study was a prospective cohort study, which did not intervene in exposure factors, but only assessed the occurrence, treatment, and prognosis of breast cancer in China.

SUMMARY:
1. To construct a prospective, multi-center breast cancer treatment cohort in China, and analyze the factors affecting breast cancer diagnosis and treatment.
2. To evaluate the diagnosis and treatment and prognosis of breast cancer among patients in different regions and hospitals.

DETAILED DESCRIPTION:
This research aims to:

A. Understand and analyze the current status of breast cancer diagnosis and treatment; B. Publish an annual report on diagnosis and treatment; C. Data sharing, dynamic evaluation; D. Evaluate consensus and guideline promotion and implementation effects; E. Propose and set clinical quality standards for industry associations, and propose improvement goals; F. Provide a basis for industry associations to formulate specialized training programs; G. To provide assistance in the formulation of health insurance policies; H. Provide a platform for clinical research on breast cancer; I. Provide evidence for the formulation of clinical guidelines and consensus

ELIGIBILITY:
Inclusion Criteria:

* Patients with malignant breast tumors must be diagnosed by cytology or histology, and their pathological types include but are not limited to breast carcinoma in situ, invasive carcinoma, and breast sarcoma.

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with malignant breast tumors
Sampling Method: Non-Probability Sample
Enrollment: 20000 (Estimated)
Dates: Start 2022-07-01 (Actual); Primary Completion 2025-07-01 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
The current status of patients diagnosed with breast cancer and their types of treatment | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 100 months
  Including but not limited to the patient receiving different surgical methods, different drugs, neoadjuvant and adjuvant therapy, etc.
Prognostic outcomes of patients | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 100 months
  Including patient disease-free survival and overall survival.

SECONDARY OUTCOMES:
Prognosis-recurrence-free survival | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 100 months
  The time from the diagnosis of breast cancer to the recurrence or metastasis of the patient, and the parts involved.
Prognosis-overall survival | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 100 months
  As the time from diagnosis of breast cancer to death of the patient

CONTACTS AND LOCATIONS:
Overall Officials: Jiong Wu, M.D, Principal Investigator — Cancer Hospital/ Institute, Fudan University
Locations (1):
- Cancer Hospital/ Institute, Fudan University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided